CLINICAL TRIAL: NCT05525494
Title: Improving Influenza Vaccination Delivery Across a Health System by the Electronic Health Records Patient Portal RCT 5
Brief Title: Patient Portal Flu Vaccine Reminders (5)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Executive Vice Chair, Vice Chair for Research, UCLA David Geffen School of Medicine, Department of Pediatrics, University of California, Los Angeles, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001889-00016; R01AI135029 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: Reminder Recall (R/R); Influenza Vaccine; Electronic Health Record; Text Message; Vaccine
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Pragmatic comparative effectiveness trial with a standard-of-care control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Text Fixed R/R Messages with Direct Appointment Schedule Link + Text Pre-Appointment Reminders (Active Comparator): Participants in this arm will receive up to 3 R/R messages by text. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment. Participants will receive a Pre-Appointment Reminder via text when they schedule a visit during the study period.
  Interventions: Behavioral: Text Fixed R/R Messages with Direct Appointment Schedule Link; Behavioral: Text Pre-Appointment Reminder
- Text Fixed R/R Messages with Direct Appointment Schedule Link (Active Comparator): Participants in this arm will receive up to 3 R/R messages by text. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Interventions: Behavioral: Text Fixed R/R Messages with Direct Appointment Schedule Link
- Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders (Active Comparator): Participants in this arm will receive a pre-commitment prompt message by portal in September. Tailored R/R messages will be sent monthly by portal based on time and place selected by patients (up to 3). R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment. Participants will receive a Pre-Appointment Reminder advising them to ask their doctor for the flu vaccine at their upcoming appointment via portal when they schedule a visit during the study period.
  Interventions: Behavioral: Portal Pre-Commitment Prompt with Tailored R/R Messages with Direct Appointment Schedule Link; Behavioral: Portal Pre-Appointment Reminder
- Portal Pre-Commitment Prompt with Tailored R/R Messages with Direct Appointment Schedule Link (Active Comparator): Participants in this arm will receive a pre-commitment prompt message by portal in September. Tailored R/R messages will be sent monthly based on time and place selected by patients (up to 3). R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Interventions: Behavioral: Portal Pre-Commitment Prompt with Tailored R/R Messages with Direct Appointment Schedule Link
- Portal Fixed R/R Messages with Direct Appointment Schedule Link + Portal Pre-Appointment Reminder (Active Comparator): Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment. Participants will receive a Pre-Appointment Reminder advising them to ask their doctor for the flu vaccine at their upcoming appointment via portal when they schedule a visit during the study period.
  Interventions: Behavioral: Portal Fixed R/R Messages with Direct Appointment Schedule Link; Behavioral: Portal Pre-Appointment Reminder
- Portal Fixed R/R Messages with Direct Appointment Schedule Link (Active Comparator): Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Interventions: Behavioral: Portal Fixed R/R Messages with Direct Appointment Schedule Link
- No R/R Message or Pre-Appointment Reminder (No Intervention): Participants do not receive any flu vaccine R/R message or Pre-Appointment Reminder advising them to ask their doctor for the flu vaccine at their upcoming appointment during the specified flu season.

INTERVENTIONS:
Behavioral: Text Fixed R/R Messages with Direct Appointment Schedule Link — Participants in this arm will receive up to 3 R/R messages by text. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Arms: Text Fixed R/R Messages with Direct Appointment Schedule Link; Text Fixed R/R Messages with Direct Appointment Schedule Link + Text Pre-Appointment Reminders
Behavioral: Text Pre-Appointment Reminder — Participants will receive a Pre-Appointment Reminder via text when they schedule a visit during the study period.
  Arms: Text Fixed R/R Messages with Direct Appointment Schedule Link + Text Pre-Appointment Reminders
Behavioral: Portal Pre-Commitment Prompt with Tailored R/R Messages with Direct Appointment Schedule Link — Participants in this arm will receive a pre-commitment prompt message by portal in September. Tailored R/R messages will be sent monthly by portal based on time and place selected by patients (up to 3). R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Arms: Portal Pre-Commitment Prompt with Tailored R/R Messages with Direct Appointment Schedule Link; Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders
Behavioral: Portal Fixed R/R Messages with Direct Appointment Schedule Link — Participants in this arm will receive up to 3 R/R messages by portal. R/R message will be sent with a Direct Appointment Scheduling link and instructions to make a flu vaccine appointment.
  Arms: Portal Fixed R/R Messages with Direct Appointment Schedule Link; Portal Fixed R/R Messages with Direct Appointment Schedule Link + Portal Pre-Appointment Reminder
Behavioral: Portal Pre-Appointment Reminder — Participants will receive a Pre-Appointment Reminder advising them to ask their doctor for the flu vaccine at their upcoming appointment via portal when they schedule a visit during the study period.
  Arms: Portal Fixed R/R Messages with Direct Appointment Schedule Link + Portal Pre-Appointment Reminder; Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders

SUMMARY:
This trial is taking place in Los Angeles, CA at clinics within the UCLA Health System.

The study design is a 2x2 nested factorial design. Patients will be randomized into 1) receiving text based reminder messages with direct scheduling link, 2) portal-based reminder messages with direct scheduling link, or 3) the control group. Patients randomized to the intervention arms will receive reminders if they are due for influenza vaccine.

Nested within the portal reminder arm, we will have two additional components for which patients will be randomized separately:

1. A pre-commitment prompt, asking patients which time (September, October, November or December) and which place (UCLA, pharmacy, workplace or school, or other) they plan to get their Influenza vaccine with tailored monthly messages based on responses (pre-commitment message with tailored recall messages with direct scheduling vs. standard portal reminders with direct scheduling).
2. A pre-appointment reminder encouraging patients to ask for their influenza vaccine at their upcoming appointment (pre-appointment reminder encouraging influenza vaccination vs. standard pre-appointment reminder not mentioning influenza vaccination)

Nested within the text message reminder arm, we will have one additional component for which patients will be randomized separately:

1) A pre-appointment reminder encouraging patients to ask for their influenza vaccine at their upcoming appointment (pre-appointment reminder encouraging influenza vaccination vs. standard pre-appointment reminder not mentioning influenza vaccination)

Despite the Advisory Committee on Immunization Practices (ACIP) recommendation in 2010 that all people above 6 months of age should receive an annual flu vaccine, vaccination rates remain low: at 6m-4.9 yrs. (70%), 5-17.9 yrs. (56%), 18-64.9 yrs. (38%), and >65 yrs. (63%). The investigators will assess the effectiveness of MyChart R/R messages and text R/R messages as compared to the standard of care control (no messages).

DETAILED DESCRIPTION:
Sub-optimal vaccination rates are a significant problem in the U.S., despite their effectiveness in preventing morbidity and mortality from vaccine-preventable illness. For influenza specifically, annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,00-80,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs.

Reminder/recall (R/R), sent by phone, mail or other modality, can improve child and adult influenza vaccination rates. However, the majority of pediatric or adult primary care practices do not conduct R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients.

A technological breakthrough that might overcome these barriers involves patient portals-- secure, web-based communication systems, embedded within electronic health records (EHRs), for patients and providers to communicate with each other via email and the internet. Portals are used by about half of Americans and half of UCLA patients. Another is text messaging at the health system level.

This randomized controlled trial will assess the effectiveness of reminders messages sent to portal users, encouraging influenza vaccination, on increasing influenza vaccination rates within a health system. Patients will be randomized into three groups: 1) one-third of patients will receive reminder messages with direct scheduling and pre-appointment reminders via the portal, 2) one-third will receive reminders via text messages with direct scheduling and pre-appointment reminders sent by the health system and 3) one-third will not receive reminders.

Patients in the portal-based reminder arm will be further randomized (separately) for two additional components: pre-commitment messages with tailored recall messages and pre-appointment reminders. Patients in the text message-based reminder arm will be further randomized for an additional component: pre-appointment reminders.

Direct scheduling: The convenience of scheduling an appointment for influenza vaccination may increase the likelihood that patients receive an influenza vaccination. All patients receiving reminders (intervention groups) will receive flu vaccine reminder letters with a link to the MyChart direct appointment scheduling page.

Pre-appointment flu reminders: Finally, a missed opportunities for vaccination occurs when patients are eligible for vaccination but are not offered a vaccine at their medical appointment. Pre-appointment reminders, sent in advance of an upcoming appointment, encouraging the patient talk to their doctor about influenza vaccination, may increase the likelihood of that patient receiving a vaccine. Patients in both the portal-based and text message-based reminder arms will be randomized to one of two groups: 1) one half will receive modified pre-appointment reminders that mention influenza vaccination and 2) one half will receive the standard pre-appointment reminders for an upcoming appointment (no mention of influenza vaccination).

Pre-commitment prompts with tailored monthly reminders: pre-planning the place and time of the flu vaccination may improve follow-through. A pre-commitment prompt will be sent via the portal in early September asking patients to commit to a time (September, October, November or December) and place (UCLA, pharmacy, workplace or school, or other) for their flu vaccination. Tailored monthly messages will be sent to patients based on their response to the pre-commitment prompt sent in September. Patients in the portal-based reminder arm will be randomized to one of two groups: 1) one half will receive the pre-commitment prompt and tailored monthly reminders, 2) one half will receive standard monthly reminders.

Interventions that apply Behavioral Economics principles in vaccine promotion messaging can increase vaccine receipt. We will include ownership language in the pre-appointment messages. The convenience of reminders sent via text and with a Direct Appointment Schedule link included enables patients to self-schedule a flu vaccine only visit, reducing friction for vaccine receipt. Additionally, the pre-commitment prompt with tailored reminders will test the principle of implementation intention (pre-planning the place and time of the flu vaccination) has been shown in other health behavior studies to improve follow-through.

For the primary analysis, the primary outcome will be the patient's end of flu season vaccination status. Intervention effects will be assessed using mixed effects log-binomial models. Models will contain terms for messaging modality (text v. portal v. none), pre-appointment reminders (sent v. not sent), and pre-commitment prompt (sent v. not sent).

The portal-based pre-commitment prompt will be sent in September of 2022. The R/R text and portal reminder messages and pre-appointment reminders and will begin in October of 2022.

ELIGIBILITY:
Inclusion Criteria:

* Active Portal Users A patient within the UCLA Health System identified as a primary care patient per an internal algorithm

Exclusion Criteria:

* A patient within the UCLA Health System not identified as a primary care patient per an internal algorithm

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 262085 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Szilagyi PG, Duru OK, Casillas A, Ong MK, Vangala S, Tseng CH, Albertin C, Humiston SG, Clark E, Ross MK, Evans SA, Sloyan M, Fox CR, Lerner C. Text vs Patient Portal Messaging to Improve Influenza Vaccination Coverage: A Health System-Wide Randomized Clinical Trial. JAMA Intern Med. 2024 May 1;184(5):519-527. doi: 10.1001/jamainternmed.2024.0001. PMID 38497955

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Fixed R/R Messages With Direct Appointment Schedule Link + Text Pre-Appointment Reminders | Text Fixed R/R Messages With Direct Appointment Schedule Link | Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders | Portal Pre-Commitment Prompt With Tailored R/R Messages With Direct Appointment Schedule Link | Portal Fixed R/R Messages With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Fixed R/R Messages With Direct Appointment Schedule Link | No R/R Message or Pre-Appointment Reminder
Started | 43682 | 43668 | 21881 | 21876 | 21864 | 21857 | 87257
Completed | 43682 | 43668 | 21881 | 21876 | 21864 | 21857 | 87257
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Fixed R/R Messages With Direct Appointment Schedule Link + Text Pre-Appointment Reminders | Text Fixed R/R Messages With Direct Appointment Schedule Link | Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders | Portal Pre-Commitment Prompt With Tailored R/R Messages With Direct Appointment Schedule Link | Portal Fixed R/R Messages With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Fixed R/R Messages With Direct Appointment Schedule Link | No R/R Message or Pre-Appointment Reminder | Total
Number analyzed (Participants) | 43682 | 43668 | 21881 | 21876 | 21864 | 21857 | 87257 | 262085
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 4096 | 4129 | 2065 | 2046 | 2028 | 2079 | 8238 | 24681
  18-64 years | 31012 | 31106 | 15587 | 15481 | 15653 | 15514 | 62084 | 186437
  65+ years | 8574 | 8433 | 4229 | 4349 | 4183 | 4264 | 16935 | 50967
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 25015 | 24820 | 12491 | 12474 | 12317 | 12420 | 49812 | 149349
  Male | 18649 | 18827 | 9378 | 9390 | 9536 | 9430 | 37418 | 112628
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown | 18 | 21 | 12 | 12 | 10 | 7 | 27 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 60 | 67 | 42 | 42 | 42 | 26 | 160 | 439
  Asian | 2739 | 2853 | 1427 | 1390 | 1381 | 1443 | 5615 | 16848
  Black | 1334 | 1357 | 654 | 652 | 704 | 651 | 2728 | 8080
  Native Hawaiian or Other Pacific Islander | 43 | 52 | 35 | 22 | 28 | 36 | 96 | 312
  White or Caucasian | 14425 | 14717 | 7286 | 7350 | 7268 | 7300 | 29118 | 87464
  Other | 4022 | 3857 | 1970 | 1887 | 1918 | 1894 | 7817 | 23365
  Multiracial | 1894 | 1981 | 978 | 972 | 1018 | 1006 | 3906 | 11755
  Unknown | 19165 | 18784 | 9489 | 9561 | 9505 | 9501 | 37817 | 113822
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5316 | 5342 | 2671 | 2662 | 2680 | 2681 | 10695 | 32047
  Not Hispanic or Latino | 31128 | 31166 | 15597 | 15639 | 15579 | 15593 | 62246 | 186948
  Unknown | 7238 | 7160 | 3613 | 3575 | 3605 | 3583 | 14316 | 43090
Primary Language [Count of Participants; unit: Participants]
  English | 42617 | 42605 | 21334 | 21282 | 21330 | 21285 | 85147 | 255600
  Spanish | 457 | 456 | 219 | 234 | 255 | 239 | 890 | 2750
  Other | 549 | 543 | 306 | 329 | 261 | 300 | 1098 | 3386
  Unknown | 59 | 64 | 22 | 31 | 18 | 33 | 122 | 349
Primary Insurance Class [Count of Participants; unit: Participants]
  Commercial | 30710 | 30719 | 15404 | 15291 | 15539 | 15391 | 61523 | 184577
  Group Health Plan | 80 | 80 | 38 | 40 | 47 | 45 | 174 | 504
  International Payor | 7 | 11 | 6 | 9 | 3 | 6 | 26 | 68
  Medi-Cal | 881 | 916 | 438 | 467 | 430 | 463 | 1869 | 5464
  Medicare | 5366 | 5376 | 2618 | 2690 | 2529 | 2686 | 10583 | 31848
  Package Billing | 0 | 2 | 0 | 1 | 2 | 0 | 3 | 8
  Tricare | 276 | 268 | 142 | 145 | 148 | 137 | 580 | 1696
  UCLA Managed Care | 5756 | 5661 | 2907 | 2919 | 2865 | 2800 | 11243 | 34151
  Other | 542 | 580 | 291 | 288 | 267 | 292 | 1120 | 3380
  Unknown | 64 | 55 | 37 | 26 | 34 | 37 | 136 | 389

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Annual Influenza Vaccine Among Index Patients
Description: Percent of patients with annual influenza vaccination (between 9/1/22 - 4/1/23) among index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/22, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Fixed R/R Messages With Direct Appointment Schedule Link + Text Pre-Appointment Reminders | Text Fixed R/R Messages With Direct Appointment Schedule Link | Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders | Portal Pre-Commitment Prompt With Tailored R/R Messages With Direct Appointment Schedule Link | Portal Fixed R/R Messages With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Fixed R/R Messages With Direct Appointment Schedule Link | No R/R Message or Pre-Appointment Reminder
Number analyzed (Participants) | 43682 | 43668 | 21881 | 21876 | 21864 | 21857 | 87257
Participants | 20689 | 20570 | 10374 | 10317 | 10369 | 10308 | 41166
Statistical Analysis 1: Comparison: Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders vs Portal Pre-Commitment Prompt With Tailored R/R Messages With Direct Appointment Schedule Link vs Portal Fixed R/R Messages With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder vs Portal Fixed R/R Messages With Direct Appointment Schedule Link vs No R/R Message or Pre-Appointment Reminder; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 0.99, 95% CI 2-sided [0.98 to 1.01] — Adjusted risk ratio. These results compare arms which received portal (any type) reminder/recall messages to the arm receiving no reminder/recall messages (control)
Statistical Analysis 2: Comparison: Text Fixed R/R Messages With Direct Appointment Schedule Link + Text Pre-Appointment Reminders vs Text Fixed R/R Messages With Direct Appointment Schedule Link vs No R/R Message or Pre-Appointment Reminder; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.00, 95% CI 2-sided [0.98 to 1.01] — Adjusted risk ratio. These results compare arms which received text (any type) reminder/recall messages to the arm receiving no reminder/recall messages (control)
Statistical Analysis 3: Comparison: Text Fixed R/R Messages With Direct Appointment Schedule Link + Text Pre-Appointment Reminders vs Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders vs Portal Fixed R/R Messages With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder vs No R/R Message or Pre-Appointment Reminder; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.01, 95% CI 2-sided [1.00 to 1.02] — Adjusted risk ratio. These results compare arms which received pre-appointment reminder/recall messages (portal and text) to the arm receiving no reminder/recall messages (control)
Statistical Analysis 4: Comparison: Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders vs Portal Pre-Commitment Prompt With Tailored R/R Messages With Direct Appointment Schedule Link vs No R/R Message or Pre-Appointment Reminder; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.00, 95% CI 2-sided [0.99 to 1.01] — Adjusted risk ratio. These results compare arms which received a tailored reminder/recall messages based on their responses to a pre-commitment questionnaire (any type) to the arm receiving no reminder/recall messages (control)

2. Primary Outcome: Number of Participants With Annual Influenza Vaccine Among Pediatric Index Patients
Description: Percent of patients with annual influenza vaccination (between 9/1/22 - 4/1/23) among pediatric index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/22, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Text Fixed R/R Messages With Direct Appointment Schedule Link + Text Pre-Appointment Reminders | Text Fixed R/R Messages With Direct Appointment Schedule Link | Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders | Portal Pre-Commitment Prompt With Tailored R/R Messages With Direct Appointment Schedule Link | Portal Fixed R/R Messages With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Fixed R/R Messages With Direct Appointment Schedule Link | No R/R Message or Pre-Appointment Reminder
Number analyzed (Participants) | 4096 | 4129 | 2065 | 2046 | 2028 | 2079 | 8238
Participants | 2132 | 2114 | 1068 | 1082 | 1090 | 1063 | 4245

ADVERSE EVENTS:
Time Frame: We did not collect information regarding adverse events.
Description: We did not collect adverse event information. We monitored whether reminder recall through the portal and text was effective at increased influenza vaccination rates. Because influenza vaccination is recommended by the Advisory Committee on Immunization Practices and is part of the U.S. recommended vaccine schedule, we did not collect adverse event data.
Arm/Group | Text Fixed R/R Messages With Direct Appointment Schedule Link + Text Pre-Appointment Reminders | Text Fixed R/R Messages With Direct Appointment Schedule Link | Portal Pre-Commitment Prompt, Tailored R/R Messages w/ Direct Scheduling + Pre-Appointment Reminders | Portal Pre-Commitment Prompt With Tailored R/R Messages With Direct Appointment Schedule Link | Portal Fixed R/R Messages With Direct Appointment Schedule Link + Portal Pre-Appointment Reminder | Portal Fixed R/R Messages With Direct Appointment Schedule Link | No R/R Message or Pre-Appointment Reminder
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT05525494/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT05525494/SAP_001.pdf